CLINICAL TRIAL: NCT06168396
Title: Testing of the Somatosensation Device (SD) for Device Effectiveness While Enhancing Feedback in Lower Extremities
Brief Title: Somatosensation Device Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Arun Jayaraman, PT, PhD, Principle Investigator, Shirley Ryan AbilityLab
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STU00219855
Record Dates: First submitted 2023-11-22; First posted 2023-12-13 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Amputation; Neuropathy
MeSH Terms: interventions — BaseLine dental cement

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline (Without Somatosensation Device) (Active Comparator): Participants will perform all outcome measures without wearing the somatosensation device.
  Interventions: Other: Baseline
- With Somatosensation Device (Experimental): Participants will perform all outcome measures while wearing the somatosensation device.
  Interventions: Device: Somatosensation Device

INTERVENTIONS:
Device: Somatosensation Device — The somatosensation device will be worn on the lower limb (either the residual limb for an amputee, or limb with decreased sensation for a participant with diabetic neuropathy) while performing outcome measures.
  Arms: With Somatosensation Device
Other: Baseline — Participants will perform outcome measures without wearing the somatosensation device.
  Arms: Baseline (Without Somatosensation Device)

SUMMARY:
This research is being done to test a new device, called the Somatosensation Device, with people who have either a below knee amputation, or neuropathy (i.e. decreased sensation) in their legs. When people have lost sensation in their feet, it may make walking and balance more difficult. The Somatosensation Device is designed to substitute the loss of feeling in a foot by pressing on nerves on the surface of the leg. It presses on the nerves by using a pneumatic balloon to put pressure on your skin. If people receive this extra sensation feedback, it may help improve their walking and balance.

ELIGIBILITY:
Inclusion Criteria:

* Have a below-knee amputation (either unilateral or bilateral) or neuropathy in their lower limbs.
* Ability to wear the somatosensation device on their lower limbs
* Ability to wear test equipment and heart rate monitors.
* Ability to follow simple directions.

Exclusion Criteria:

* History of severe back pain in the last 3 months.
* History of severe knee pain in the last 3 months.
* Unable to walk for 3 minutes with or without an assistive device
* Poor skin integrity (i.e open wounds, skin breakdown) that could be made worse by wearing the somatosensation device.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Functional Gait Assessment (FGA) | Baseline, during the intervention
  The Functional Gait Assessment is a test to assess an individual's postural stability and ability to perform multiple motor tasks while walking. Tests include walking at different speeds, walking with head turns, turns, stepping over obstacles, walking tandem, walking with eyes closed, walking backwards, and stair navigation. Scores are on a 0-30 scale, with higher scores showing better balance and mobility.

SECONDARY OUTCOMES:
10 Meter Walk Test | Baseline, during the intervention
  The 10MWT assesses walking speed in meters per second. In the 10MWT, subjects are directed to walk at their self-selected and maximum safe speed with the effects of acceleration and deceleration minimized (by adding 2 meters at the beginning and at the end of the course to isolate the subject's steady state speed). Any assistive device and orthotic should be kept consistent and documented. Participants will complete three trials at their self-selected speed and three trials at their fast but still safe speed. This will be performed over the GAITRite electronic walkway, to measure temporal-spatial gait parameters.
Mini-BESTest | Baseline, during the intervention
  A multi-task balance assessment that identifies postural control problems across a wide variety of situations.
Activities Specific Balance Confidence Scale (ABC) | Baseline, during the intervention
  A self-reported questionnaire that measures a participant's confidence in their balance in performing various activities without falling or becoming unsteady. Scores are on a 0-100% confidence scale, with higher scores equaling greater confidence.
Vestibular Disorders Activities of Daily Living Scale (VADL) | Baseline, during the intervention
  A self-reported questionnaire that evaluates the effects of vertigo and balance disorders on independence routine activities of daily living. Scores range from 1-8, with lower scores indicating greater independence with activities.

CONTACTS AND LOCATIONS:
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States